CLINICAL TRIAL: NCT01498471
Title: NICE Guideline 'Red Flags' to Predict Serious Outcome After Transient Loss of Consciousness: Prospective Validation Study in the Emergency Department.
Brief Title: NICE Guideline 'Red Flags' to Predict Serious Outcome After Transient Loss of Consciousness
Status: Withdrawn | Type: Observational
Why Stopped: longterm abscence of investigator
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: UZ/PVB/2011
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study is designed to evaluate the accuracy of the National Institute for Health and Clinical Excellence (NICE) guideline 'red flags' to identify patients at high risk of short term serious outcome when presenting in the emergency department (ED) with Transient Loss of Consciousness (TLoC). Red flags were defined as ECG abnormality, history or physical signs of heart failure, TLoC during exercise, family history of sudden cardiac death at an age < 40 years and/or an inherited cardiac condition, new or unexplained breathlessness, heart murmur, absence of prodromal symptoms in any patient aged > 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>= 16 years) with a complaint of TLoC

Exclusion Criteria:

* Patients needing immediate treatment, with trauma related or drug or alcohol related TLoC were excluded, as well as patient with persistent altered level of consciousness, simple fall and drop attack

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients (>= 16 years) presenting in the ED with a complaint of TLoC
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
serious outcome | day 7
  death, myocardial infarction, arrhythmias, pulmonary embolism, stroke or transient ischemic attack, subarachnoid or non traumatic cerebral haemorrhage, aortic dissection, new diagnosis of structural heart disease thought to be related to syncope, and significant haemorraghe or anemia requiring blood transfusion, readmission for similar symptoms related to the initial event and acute intervention during hospital admission

SECONDARY OUTCOMES:
serious outcome | 1 year
  death, myocardial infarction, arrhythmias, pulmonary embolism, stroke or transient ischemic attack, subarachnoid or non traumatic cerebral haemorrhage, aortic dissection, new diagnosis of structural heart disease thought to be related to syncope, and significant haemorraghe or anemia requiring blood transfusion, readmission for similar symptoms related to the initial event and acute intervention during hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- See also: Related Info — http://www.nice.org.uk/guidance/CG109